CLINICAL TRIAL: NCT06267690
Title: Development and Validation of a CT-based Radiomics Model to Predict Survival-graded Fibrosis in Pancreatic Ductal Adenocarcinoma
Brief Title: A CT-based Radiomics Model to Predict Survival-graded Fibrosis in PDAC
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Siya Shi, clinical doctor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: SYSUFAH2021025
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tumor tissue specimens were fixed in 10% formalin and processed routinely. The tumor area with the richest fibrosis was selected, sectioned at a thickness of 4 μm, and stained using Masson's trichrome stain. The collagen fraction (CF), a quantitative substitute for fibrosis, was analyzed using ImageJ software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high fibrosis group: No intervention had been adminstered during treatment of patients.
  Interventions: Procedure: surgery
- low fibrosis group: No intervention had been adminstered during treatment of patients.
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — Patients with suspected pancreatic cancer who underwent contrast-enhanced CT and pathological examinations after the surgery.

SUMMARY:
Tumor fibrosis plays an important role in chemotherapy resistance in pancreatic ductal adenocarcinoma (PDAC), however there remains a contradiction in the prognostic value of fibrosis. We aimed to investigate the relationship between tumor fibrosis and survival in patients with PDAC, classify patients into high- and low-fibrosis groups, and develop and validate a CT-based radiomics model to non-invasively predict fibrosis before treatment.

DETAILED DESCRIPTION:
This retrospective, bicentric study included 295 pretreated patients with PDAC. Tumor fibrosis was assessed using the collagen fraction (CF). Clinical-pathological variables were gathered, and radiological features were evaluated by three radiologists in consensus. The patients were followed up at 1, 3, 6, and 9 months postoperatively and every 3-6 months thereafter. All follow-up examinations included carbohydrate antigen 19-9 (CA 19-9) measurements and imaging (contrast-enhanced CT, contrast-enhanced MRI, ultrasonography, or positron emission tomography). The overall survival (OS) and disease-free survival (DFS) were also recorded. Cox regression analysis was used to evaluate the associations of CF with OS and DFS. Receiver operating characteristic (ROC) analyses were used to determine the rounded threshold of CF. An integrated model (IM) was developed by incorporating selected radiomic features and clinical-radiological characteristics. The predictive performance was validated in the test cohort (Center 2). It was hypothesized that tumor fibrosis could be classified into two survival-graded groups and that the incorporation of radiomics features and clinical-radiological features would help predict the status of fibrosis. Thus, the association between fibrosis and overall survival (OS)/disease-free survival (DFS) was determined, and the patients with PDAC were divided into high- and low-CF groups in this study. In addition, a CT-based radiomics model was developed and validated to non-invasively predict fibrosis before treatment in patients with PDAC from two centers. It was hypothesized that the performance of the integrated model would be superior to that of the clinical-radiological model.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected pancreatic tumors who underwent contrast-enhanced CT and pathological examinations at Center 1 and Center 2 were eligible for inclusion in this study.

Exclusion Criteria:

* (a) pathologically diagnosed PDAC by resection; (b) time intervals between contrast-enhanced CT and pathology less than 2 weeks; (c) no history of previous treatment such as resection, chemotherapy, or radiotherapy. The patients were excluded as follows: (a) unavailable pathological sections for evaluating the fibrosis; (b) incomplete clinical records; (c) missing CT images or poor CT image quality; (d) coincidence of other malignant tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected pancreatic tumors who underwent contrast-enhanced CT and pathological examinations at Center 1 and Center 2 were eligible for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
fibrosis | after the surgery
  percentage

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Ting Feng, MD, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Shi Siya, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
All data generated for this study are from the corresponding author upon reasonable request.